CLINICAL TRIAL: NCT01155661
Title: Long-Term, Open-Label, Safety Study of LY2216684 12 to 18 mg Once Daily as Adjunctive Treatment for Patients With Major Depressive Disorder Who Are Partial Responders to Selective Serotonin Reuptake Inhibitor Treatment
Brief Title: A Safety Study in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11318; H9P-MC-LNBO (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2216684 (edivoxetine) + SSRI (Experimental)
  Interventions: Drug: LY2216684 (edivoxetine); Drug: SSRI

INTERVENTIONS:
Drug: LY2216684 (edivoxetine) — 12 to 18 milligrams (mg), administered orally, once daily for 54 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Other Names: LY2216684; edivoxetine
Drug: SSRI — Participants should have been on their SSRI for at least 6 weeks prior and were to continue on their stable dose throughout the study.
  Other Names: Selective Serotonin Reuptake Inhibitor

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of LY2216684 administered once daily (QD) in the adjunctive treatment with a selective serotonin reuptake inhibitor (SSRI) for up to approximately 1 year in participants with major depressive disorder (MDD) who are partial responders to their SSRI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults competent and able to give informed consent
* Women of child-bearing potential may participate but must test negative for pregnancy at the time of study entry; both women/men agree to use a reliable method of birth control
* Participants who are being treated with one of the following selective serotonin reuptake inhibitors (SSRIs): escitalopram, citalopram, sertraline, fluoxetine, paroxetine, and fluvoxamine; for at least 6 weeks prior to investigational product dispensing with at least the last 4 weeks at a stable, optimized dose
* Drug and dosage should be within the labeling guidelines for the specific country
* Meet criteria for Major Depressive Disorder (MDD), as defined by the Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR) criteria
* Meet criteria for partial response, as defined by investigator's opinion that participant has experienced a minimal clinically meaningful improvement with SSRI
* Have a Grid Hamilton Rating Scale for Depression (GRID-HAMD17) total score greater than or equal to 16 at screening
* Have less than or equal to 75 percent improvement on the current SSRI at screening determined by the Massachusetts General Hospital Antidepressant Response Questionnaire (MGH-ATRQ)
* Meet all other inclusion criteria per protocol

Exclusion Criteria:

* Presence of another primary psychiatric illnesses:

  * Have had or currently have any additional ongoing DSM-IV-TR Axis I condition other than major depression within 1 year of screening
  * Have had any anxiety disorder that was considered a primary diagnosis within the past year (including panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, and social phobia, but excluding specific phobias)
  * Have a current or previous diagnosis of a bipolar disorder, schizophrenia, or other psychotic disorder
  * Have a history of substance abuse and/or dependence within the past 1 year (drug categories defined by DSM-IV-TR), not including caffeine and nicotine
  * Have a DSM-IV-TR Axis II disorder that, in the judgment of the investigator, would interfere with compliance with protocol
* Unstable medical conditions that contraindicate the use of LY2216684

  * Have any diagnosed medical condition which could be exacerbated by noradrenergic agents including unstable hypertension, unstable heart disease, tachycardia, tachyarrhythmia, narrow-angled glaucoma, urinary hesitation or retention
* Use of excluded concomitant or psychotropic medication other than SSRI
* Have initiated or discontinued hormone therapy within the previous 3 months of prior to enrollment
* History of treatment resistant depression as shown by:

  * Have had lack of response of the current depressive episode to 2 or more adequate courses of antidepressant therapy at a clinically appropriate dose for at least 4 weeks, or in the judgment of the investigator, the participant has treatment-resistant depression
  * Have a history of electroconvulsive therapy, transcranial magnetic stimulation, or psychosurgery within the last year
* Meet any other exclusion criteria per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (48):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cerritos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Alamitos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redlands, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Walton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Princeton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Kisco, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Brazil (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aparecida de Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belo Horizonte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Botucatu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pelotas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ribeirão Preto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salvador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Chile (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antofagasta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago
- Lithuania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipėda
- Mexico (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., León
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mazatlán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villahermosa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zapopan
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heerde
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildervank
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcalá de Henares
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zamora

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a 54 week LY2216684 treatment Open-label Phase followed by 1 week Discontinuation Phase after abrupt discontinuation of treatment.
Groups:
- LY2216684 + SSRI: LY2216684 (edivoxetine): 12 to 18 milligrams (mg), administered orally, once daily for 54 weeks, adjunctive to selective serotonin reuptake inhibitor (SSRI)
Period: Overall Study
Arm/Group | LY2216684 + SSRI
Started | 608
Completed | 328
Not Completed | 280
Not completed — Adverse Event | 101
Not completed — Death | 1
Not completed — Lack of Efficacy | 32
Not completed — Lost to Follow-up | 22
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 35
Not completed — Withdrawal by Subject | 73
Not completed — Sponsor Decision | 13

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 608
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.54 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455
  Male | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 214
  Not Hispanic or Latino | 320
  Unknown or Not Reported | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 59
  White | 521
  More than one race | 9
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 300
  Mexico | 110
  Brazil | 82
  Chile | 50
  Lithuania | 38
  Netherlands | 19
  Spain | 9

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Clinically Significant Effects
Description: A clinically significant effect was defined as a serious adverse event, regardless of causality.
  A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through 54 weeks
Population: All enrolled participants who did not discontinue from the study for the reason 'Lost to follow-up' at the first post-baseline visit.
Measure: Number; unit: participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 600
participants | 13

2. Secondary Outcome: Percent of Participants With Suicidal Ideation and Behavior Based on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation was defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which included a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide.
Time Frame: Baseline through Week 54
Population: All enrolled participants with a baseline and at least one post-baseline C-SSRS value.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 589
percentage of participants
  Suicidal Ideation | 11.71
  Suicidal Behavior | 0.17

3. Secondary Outcome: Change From Baseline to 54 Week Endpoint in the Arizona Sexual Experiences (ASEX) Scale
Description: The ASEX scale was used to assess sexual functioning in both males and females. The ASEX total score for the male and female version was calculated as the sum of the responses (rated from 1 [extremely] to 6 [no/never]) to the 5 items of the ASEX scale. Total scores ranged from 5 to 30 with higher scores indicating greater sexual dysfunction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline ASEX total score value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 537
units on a scale | -2.28 (0.25)

4. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ)
Description: The CPFQ is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item was scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total scores ranged from 7 to 42. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline CPFQ total score value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 541
units on a scale | -8.64 (0.30)

5. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score and Individual Items
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline MADRS individual item and total score value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 589
units on a scale
  MADRS Item 1: Apparent Sadness | -2.17 (0.05)
  MADRS Item 2: Reported Sadness | -2.38 (0.06)
  MADRS Item 3: Inner Tension | -1.56 (0.06)
  MADRS Item 4: Reduced Sleep | -1.97 (0.07)
  MADRS Item 5: Reduced Appetite | -1.08 (0.04)
  MADRS Item 6: Concentration Difficulties | -1.88 (0.06)
  MADRS Item 7: Lassitude | -2.18 (0.06)
  MADRS Item 8: Inability to Feel | -2.22 (0.06)
  MADRS Item 9: Pessimistic Thoughts | -1.52 (0.05)
  MADRS Item 10: Suicidal Thoughts | -0.26 (0.02)
  MADRS Total Score | -16.97 (0.41)

6. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression subscales. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.' Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Hospital Anxiety and Depression Scale (HADS) depression subscale value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 588
units on a scale | -6.32 (0.21)

7. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Clinical Global Impression - Severity (CGI-S)
Description: Clinical Global Impression - Severity (CGI-S) measures severity of depression at the time of assessment compared with the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Clinical Global Impression - Severity (CGI-S) value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 589
units on a scale | -2.17 (0.06)

8. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Fatigue Associated With Depression (FAsD) Average Score and Subscale Scores
Description: The Fatigue Associated with Depression (FAsD) is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The "Experience Score" was derived by taking the mean of Items 1 through 6, the "Impact Score" was derived by taking the mean of Items 7 through 13 (applicable items only), and the "Average Score" was the mean of Items 1 through 13 (derived by taking the mean of all applicable items for each participant). Item 12 applied only to participants with a spouse or significant other and Item 13 applied to participants who had a job or who went to school. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Fatigue Associated with Depression (FAsD) average score and subscale score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 541
units on a scale
  FAsD Experience Score | -1.25 (0.05)
  FAsD Impact Score | -1.37 (0.05)
  FAsD Average Score | -1.30 (0.05)

9. Secondary Outcome: Probability of Meeting the Response Criteria for Depressive Symptoms at Week 54 Endpoint
Description: Response criteria was defined as at least a 50% decrease from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) total score. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). This analysis models the probability of response at each visit, and the estimated probabilities were adjusted for visit and the baseline MADRS total score.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Montgomery-Asberg Depression Rating Scale (MADRS) total score value.
Measure: Number; unit: Probability of response
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 589
Probability of response | 0.772 (0.020)

10. Secondary Outcome: Probability of Meeting the Remission Criteria for Depressive Symptoms at Week 54 Endpoint
Description: Remission criteria was defined as a Montgomery-Asberg Depression Rating Scale (MADRS) total score of <= 10. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). This analysis models the probability of remission at each visit, and the estimated probabilities were adjusted for visit and the baseline MADRS total score.
Time Frame: Baseline, Week 54
Population: as for outcome 9
Measure: Number; unit: Probability of remission
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 589
Probability of remission | 0.758 (0.022)

11. Secondary Outcome: Percentage of Participants Who Meet Response Criteria of Depressive Symptoms by Week 8
Description: Response criteria was defined as at least a 50% decrease from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) total score. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). The Kaplan-Meier product limit method of time to first response was calculated. In the calculation, participants who did not meet response criteria were considered as right-censored observations. The estimated percentage of participants who met response criteria by Week 8 from the Kaplan-Meier method is presented.
Time Frame: Baseline, Week 8
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 589
percentage of participants | 59.2

12. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale Score
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item was rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression subscale. Scores of 11 or more on either subscale were considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.' Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Hospital Anxiety and Depression Scale (HADS) anxiety subscale value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 588
units on a scale | -4.57 (0.18)

13. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Sheehan Disability Scale (SDS) Total Score and Subscores
Description: The Sheehan Disability Scale (SDS) Global Functional Impairment Score (total score) and Subscores were completed by the participant and were used to assess the effect of the participant's symptoms on their work (Item 1), social (Item 2), and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. The Global Functional Impairment Score is the sum of the 3 items, and scores ranged from 0 to 30 with higher values indicating greater disruption in the participant's work life (work/school impairment [imp] score), social life (social life/leisure activities impairment [imp] score), and family life (family life/home responsibilities impairment [imp] score). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Sheehan Disability Scale (SDS) subscale score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 491
units on a scale
  SDS Global Functional Impairment(Imp) Score: number analyzed (Participants) | 490
  SDS Global Functional Impairment(Imp) Score | -10.71 (0.37)
  Work/School Imp Score: number analyzed (Participants) | 318
  Work/School Imp Score | -3.36 (0.15)
  Social Life/Leisure Activity Imp Score | -3.74 (0.13)
  Family Life/Home Responsibility Imp Score: number analyzed (Participants) | 490
  Family Life/Home Responsibility Imp Score | -3.61 (0.13)

14. Secondary Outcome: Change From Baseline to 54 Week Endpoint in EuroQol Questionnaire - 5 Dimension (EQ-5D)
Description: The EQ-5D Visual Analog Scale is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score is self-reported using a visual analogue scale, marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline EuroQol Questionnaire - 5 Dimension (EQ-5D) visual analog scale value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 488
units on a scale | 23.607 (1.019)

15. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) is a self-administered 16 item questionnaire measuring degree of enjoyment and satisfaction experienced in various areas of daily life during the past week on a 5-point Likert scale (1=very poor and 5=very good). The total raw score is the sum of Items 1 to 14 and ranges from 14 to 70. The raw scores are converted to and expressed as the percentage of the maximum possible score. Higher scores indicate higher levels of enjoyment/satisfaction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline score, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) percent of maximum possible score value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 491
units on a scale | 21.56 (0.90)

16. Secondary Outcome: Percentage of Participants Who Reported Resource Utilization (RU) at Baseline and at the Week 54 Endpoint
Description: The Resource Utilization (RU) form assesses the frequency and type of medical services (a primary care visit and/or a psychiatrist visit) that participants used within the previous year (for the baseline visit) or within approximately the previous 3 months (for post-baseline visits or the Week 54 endpoint). The percentage of participants who reported greater than zero number of primary care doctor visits and greater than zero number of psychiatrist visits is presented.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline Resource Utilization value.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 607
percentage of participants
  Primary Care Doctor Visits, Baseline | 62.27
  Primary Care Doctor Visits, Week 54: number analyzed (Participants) | 338
  Primary Care Doctor Visits, Week 54 | 30.18
  Psychiatrist Visits, Baseline | 44.15
  Psychiatrist Visits, Week 54: number analyzed (Participants) | 337
  Psychiatrist Visits, Week 54 | 4.75

17. Secondary Outcome: Percentage of Participants With Discontinuation-Emergent Adverse Events (DEAEs)
Description: Discontinuation-emergent adverse events (DEAEs) were events that first occurred or worsened within 1-week after abrupt discontinuation of LY2216684 (edivoxetine) treatment.
Time Frame: Up to1 week after discontinuation of treatment
Population: All enrolled participants who abruptly discontinued LY2216684 (edivoxetine) treatment either at the end of the study or after early withdrawal from the study and who did not discontinue from the study for the reason 'Lost to follow-up' at the first post-baseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 472
percentage of participants | 20.97

18. Secondary Outcome: Percentage of Participants Who Meet Remission Criteria of Depressive Symptoms by Week 8
Description: Remission criteria was defined as a Montgomery-Asberg Depression Rating Scale (MADRS) total score of <= 10. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). The Kaplan-Meier product limit method of time to first remission was calculated. In the calculation, participants who did not meet remission criteria were considered as right-censored observations. The estimated percentage of participants who meet remission criteria by Week 8 from the Kaplan-Meier method is presented.
Time Frame: Baseline, Week 8
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 589
percentage of participants | 47.7

19. Secondary Outcome: Plasma Concentration of LY2216684
Time Frame: Weeks 2, 6, and 8
Population: All enrolled participants with at least one plasma sample.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2216684 + SSRI: LY2216684: 12 to 18 milligrams (mg), administered orally, once daily for 54 weeks, adjunctive to selective serotonin reuptake inhibitor (SSRI)
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 512
nanograms per milliliter (ng/mL)
  12 mg dose: number analyzed (Participants) | 496
  12 mg dose | 29.6 (21.4)
  18 mg dose: number analyzed (Participants) | 262
  18 mg dose | 53.6 (35.7)

20. Secondary Outcome: The Number of Participants Experiencing Clinically Significant Effects as a Function of CYP2D6 Predicted Phenotype at Week 54 Endpoint
Description: A clinically significant effect was defined as a treatment-emergent adverse event; a reported adverse event that first occurred or worsened during the treatment phase. CYP2D6 predicted phenotype was classified as poor metabolizer (PM) or non-poor metabolizer (non-PM). The number of participants who reported at least one treatment-emergent adverse event is presented for each phenotype classification.
Time Frame: Baseline, Week 54
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 600
participants
  Poor Metabolizer: number analyzed (Participants) | 22
  Poor Metabolizer | 17
  Non-poor Metabolizer: number analyzed (Participants) | 539
  Non-poor Metabolizer | 408

21. Secondary Outcome: Change From Baseline to 54 Week Endpoint in Blood Pressure
Description: Blood pressure measurements were collected when the participant was in a sitting position. Three measurements of sitting blood pressure collected at approximately 1-minute intervals at every visit were averaged and used as the value for the visit. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline value, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline blood pressure value.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mm Hg)
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 590
millimeters of mercury (mm Hg)
  Sitting Systolic Blood Pressure | 2.28 (0.50)
  Sitting Diastolic Blood Pressure | 2.17 (0.40)

22. Secondary Outcome: Change From Baseline to Week 54 Endpoint in Pulse Rate
Description: Pulse measurements were collected when the participant was in a sitting position. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for investigator, visit, baseline value, and baseline-by-visit.
Time Frame: Baseline, Week 54
Population: All enrolled participants with a baseline and at least one post-baseline pulse rate value.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 590
beats per minute (bpm) | 7.01 (0.49)

ADVERSE EVENTS:
Groups:
- LY2216684 + SSRI Open-Label Phase: LY2216684 (edivoxetine): 12 to 18 milligrams (mg), administered orally, once daily for 54 weeks, adjunctive to selective serotonin reuptake inhibitor (SSRI); included all enrolled participants who did not discontinue from the study for the reason 'Lost to follow-up' at the first post-baseline visit.
- Discontinuation Phase: Included all enrolled participants who abruptly discontinued LY2216684 (edivoxetine) treatment either at the end of the study or after early withdrawal from the study and who did not discontinue from the study for the reason 'Lost to follow-up' at the discontinuation phase visit. All participants maintained their SSRI treatment at the stable dose during the discontinuation phase.
Arm/Group | LY2216684 + SSRI Open-Label Phase | Discontinuation Phase
Serious Adverse Events (participants affected / at risk) | 13/600 | 0/472
Other Adverse Events (participants affected / at risk) | 448/600 | 99/472
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 + SSRI Open-Label Phase (N=600) | Discontinuation Phase (N=472)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — resulted in death
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Bartholinitis (Reproductive system and breast disorders) | 1/452 (1) | 0/362 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 + SSRI Open-Label Phase (N=600) | Discontinuation Phase (N=472)
Palpitations (Cardiac disorders) | 25 (26) | 4 (4)
Constipation (Gastrointestinal disorders) | 72 (77) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 56 (58) | 2 (2)
Nausea (Gastrointestinal disorders) | 88 (99) | 12 (12)
Vomiting (Gastrointestinal disorders) | 40 (46) | 1 (1)
Chills (General disorders) | 21 (23) | 0 (0)
Influenza (Infections and infestations) | 21 (25) | 3 (3)
Nasopharyngitis (Infections and infestations) | 19 (22) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 34 (39) | 0 (0)
Dizziness (Nervous system disorders) | 45 (50) | 15 (18)
Headache (Nervous system disorders) | 68 (107) | 51 (59)
Somnolence (Nervous system disorders) | 21 (26) | 7 (7)
Anxiety (Psychiatric disorders) | 20 (23) | 7 (7)
Insomnia (Psychiatric disorders) | 36 (38) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 7/148 (7) | 0/110 (0)
Testicular pain (Reproductive system and breast disorders) | 5/148 (5) | 0/110 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 85 (93) | 3 (3)
Hypertension (Vascular disorders) | 23 (25) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days